CLINICAL TRIAL: NCT05042401
Title: Safety, Tolerability, and Pharmacokinetics/Pharmacodynamics of a Single Subcutaneous Injection of SHR-1703 in Patients With Asthma -- a Randomized, Double-blind, Dose-increasing, Placebo Controlled Phase I Clinical Study
Brief Title: A Trial of SHR-1703 in Asthma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1703-103
Record Dates: First submitted 2021-07-20; First posted 2021-09-13 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2022-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: SHR-1703 low dose VS. placebo low dose. SHR-1703 high dose VS. placebo high dose
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment group A (Experimental)
  Interventions: Drug: SHR-1703
- Treatment group B (Placebo Comparator)
  Interventions: Drug: placebo
- Treatment group C (Experimental)
  Interventions: Drug: SHR-1703
- Treatment group D (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: SHR-1703 — SHR-1703 low dose
  Arms: Treatment group A
Drug: placebo — placebo low dose
  Arms: Treatment group B
Drug: SHR-1703 — SHR-1703 high dose
  Arms: Treatment group C
Drug: placebo — placebo high dose
  Arms: Treatment group D

SUMMARY:
SHR-1703 is a monoclonal antibody under development for severe asthma. This study is the first study in patients with asthma. The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics ，pharmacodynamics and immunogenic characteristics of multiple subcutaneous injections of SHR-1703 in asthmatic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
2. Able to read, comprehend and write at a sufficient level to complete study materials.
3. Aged 18 to 65 years (inclusive).
4. Body weight equal or more than 40.0 kg.
5. Diagnosis of asthma
6. The condition was stable 4 weeks before screening, and no drugs or standard asthma drugs were used. Treatment medications include asthma maintenance medications and/or emergency relief medications as needed. If the use of asthma maintenance treatment drugs, it is necessary to maintain a stable usage and dosage and stable condition. Asthma maintenance medications include one or more of inhaled corticosteroids (ICS), inhaled long-acting beta2 agonists (LABA), and inhaled long-acting cholinergic receptor antagonists (LAMA). Emergency relief drugs are limited to short-acting β2 receptor agonists (SABA) or short-acting cholinergic receptor antagonists (SAMA) inhaled on demand;
7. Serum eosinophil count at screening and baseline ≥0.15/L;
8. Alanine aminotransferase (ALT), aspartate aminotransferase (AST) and total bilirubin were less than the upper limit of normal range (ULN) during screening;
9. During the screening period, the FEV1/ estimated value of lung function test before bronchodilators was ≥45% (the examination time was between 6:00 a.m. and 12:00 a.m.), and the short-acting bronchodilators were stopped for at least 4 hours before the examination;
10. Subjects (including partners) had no family planning and were voluntarily using effective contraceptives during the study period and during the last visit (see appendix for specific contraceptives).

Exclusion Criteria:

1. People who are allergic to IL-5 antibody drugs and excipients or other biological agents;
2. Patients with diseases other than asthma that lead to elevated blood eosinophilic granulomatosis, including but not limited to eosinophilic granulomatosis with polyangiitis (EGPA), eosinophilic esophagitis, etc.;
3. Have a history or history of clinically significant lung diseases other than asthma, including active pulmonary tuberculosis, bronchiectasis, pulmonary fibrosis, bronchopulmonary aspergillosis, chronic obstructive pulmonary disease, lung cancer, etc.;
4. ≥1 clinically significant exacerbation of asthma within 4 weeks prior to screening or within the screening period (clinically significant exacerbation of asthma was defined as ≥3 days of systemic glucocorticosteroid treatment and/or exacerbation of asthma requiring emergency department visits and hospitalization);
5. A life-threatening acute exacerbation of asthma occurred within 5 years prior to screening. Acute episodes of life-threatening asthma were defined as requiring intubation and/or hypercapnia, respiratory arrest or disturbance of consciousness;
6. Bacterial or viral infection of the upper or lower respiratory tract, sinus, or middle ear, occurring within 4 weeks prior to baseline, resulting in changes in asthma management or, in the investigator's opinion, possible changes that are expected to affect subjects' asthma status or their ability to participate in the study;
7. Patients with a history of malignant tumor;
8. The combination of other disease states and/or medical interventions that interfere with clinical research. Interference with clinical studies includes but is not limited to interference with liver and kidney function and other safety data analysis, blood eosinophil level analysis, etc
9. Hepatitis B virus surface antigen (HBsAg), human immunodeficiency virus antibody (HIV-AB), syphilis serological test, hepatitis C virus antibody (HCV-AB) were positive during screening;
10. Participants in any drug clinical trial within 3 months prior to baseline were defined as: participants in the trial drug (excluding placebo); Or they are still in the follow-up period of a clinical study or within the 5 half-life of the investigational drug, whichever is longer, before screening;
11. Received any biologic treatment for inflammatory disease in the 6 months prior to baseline that affected asthma and/or blood eosinophil levels, or did not exceed 5 half-lives, whichever is longer;
12. Regular systemic use of glucocorticoids for conditions other than asthma during the 6 months prior to baseline;
13. Before using the study drug use within 14 days of any interference on clinical studies (including but not limited to affect kidney function, blood eosinophil level, etc.) of drugs (including prescription drugs, over-the-counter drugs, Chinese herbal medicine and dietary supplements, etc.), or use of drugs is not more than five half-life of longer (in); Prescription drugs include but are not limited to: Penicillin and cephalosporin, sulfa, tetracycline, granulocyte macrophage colony stimulating factor (gm-csf), interleukin 2 (IL 2) and ranitidine non-steroidal anti-inflammatory drugs, ureide within, allopurinol, b, L - tryptophan, willow nitrogen sulfonyl pyridine, carbamazepine, hydrochlorothiazide, ring spore, nevirapine, clozapine, o o n peace made pp azole, etc .
14. Blood donation history within 1 month before screening, or severe blood loss (total blood volume ≥400 mL), or received blood transfusion within 2 months;
15. Those who receive live (attenuated) vaccine within 1 month prior to screening or plan to receive live (attenuated) vaccine during the test;
16. Suspected parasitic infection/infection within 6 months prior to screening;
17. Pregnancy status (defined as a state from conception to termination of pregnancy and positive for human chorionic gonadotropin) or breastfeeding;
18. Previous smokers who had smoked for 6 months prior to screening or who had quit smoking for more than 6 months at the time of screening had smoked more than 10 pack-years (pack-years = number of years of smoking × number of packs per day). Alcohol consumption within 3 months prior to screening (average consumption of ≥14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of spirits, or 100 m1 of wine). Have a history of substance abuse within 5 years;
19. Positive smoke screen, drug screen and alcohol breath test during screening;
20. Researchers and related staff of the research center or others directly involved in the implementation of the program;
21. The investigator considers that there are any other factors that may cause the subject to fail to complete the study or present a significant risk to the subject.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2023-06-15 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
The incidence of adverse events of SHR-1703 | From Day 1 to Day 281
Severity of adverse events of SHR-1703 | From Day 1 to Day 281
Tolerability of adverse events of SHR-1703 | From Day 1 to Day 281

SECONDARY OUTCOMES:
Evaluate the concentrations of multiple subcutaneous injections of SHR-1703 in asthmatic patients | From Day 1 to Day 281
The percentage change of absolute eosinophil count from baseline | From Day 1 to Day 281
Incidence of SHR-1703 immunogenicity | From Day 1 to Day 281
Occurrence time of SHR-1703 immunogenicity | From Day 1 to Day 281
Duration of anti drug antibody (ADA) of SHR-1703 | From Day 1 to Day 281
Titer of anti drug antibody (ADA) of SHR-1703 | From Day 1 to Day 281
The percentage change of forced expiratory volume in 1 second from baseline | From Day 1 to Day 281
The percentage change of forced vital capacity from baseline | From Day 1 to Day 281

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided